CLINICAL TRIAL: NCT00907348
Title: Prospective Multicenter Dose Finding Phase II Pilot Trial to Evaluate Efficacy and Safety of Treatment With Lenalidomide Plus R-CHOP21 (LR-CHOP21) for Elderly Patients With Untreated Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: Prospective Multicenter Dose Finding Phase II Pilot Trial to Evaluate Efficacy and Safety of LR-CHOP21 for Elderly Patients With Untreated Diffuse Large B Cell Lymphoma
Acronym: REAL07
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIL_REAL07
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Non Hodgkin Lymphoma; Follicular Lymphoma
Keywords: NHL; Non Hodgkin Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohorts 1 - 2 - 3 - 4 (Experimental): Chemiotherapy
  Interventions: Drug: LR-CHOP21

INTERVENTIONS:
Drug: LR-CHOP21 — FIRST DOSE LEVEL: Rituximab 375 mg/sqm D 0 or 1; Cyclophosphamide 750 mg/sqm iv D1; Doxorubicin 50 mg/sqm iv D1; Vincristine 1.4 mg/sqm iv D1; Prednisone 40 mg/sqm orally D1, D2, D3, D4, D5; Revlimid 5 mg/day D1-D14
  SECOND DOSE LEVEL: Rituximab 375 mg/sqm D 0 or 1;Cyclophosphamide 750 mg/sqm iv D1; Doxorubicin 50 mg/sqm iv D1; Vincristine 1.4 mg/sqm iv D1; Prednisone 40 mg/sqm orally D1, D2, D3, D4, D5; Revlimid 10 mg/day D1-D14
  THIRD DOSE LEVEL: Rituximab 375 mg/sqm D 0 or 1; Cyclophosphamide 750 mg/sqm iv D1; Doxorubicin 50 mg/sqm iv D1; Vincristine 1.4 mg/sqm iv D1; Prednisone 40 mg/sqm orally D1, D2, D3, D4, D5; Revlimid 15 mg/day D1-D14
  FOURTH DOSE LEVEL: Rituximab 375 mg/sqm D 0 or 1; Cyclophosphamide 750 mg/sqm iv D1; Doxorubicin 50 mg/sqm iv D1; Vincristine 1.4 mg/sqm iv D1; Prednisone 40 mg/sqm orally D1, D2, D3, D4, D5; Revlimid 20 mg/day D1-D14 Repeated every 21 days

SUMMARY:
This is a prospective multicenter phase II pilot trial designed with the purpose of dose finding to evaluate the efficacy and safety of treatment with Lenalidomide plus R-CHOP21 (LR-CHOP21) for elderly patients with untreated Diffuse Large B Cell Lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form
2. Able to adhere to the study visit schedule and other protocol requirements
3. Histologic subtypes as follows:

   * CD20 positive Diffuse large B-Cell lymphoma
   * CD20 positive Follicular grade IIIb
4. Age 60-80
5. Untreated patients. In patients with bulky mass or systemic symptoms or compressive disease or rapidly progressive adenopathies a pre-study treatment is allowed with steroids and/or a single dose of Vincristine 1.4 mg/mq (max 2) in the seven days prior the start of the study treatment
6. Measurable and/or evaluable disease
7. Ann Arbor stage II, III, IV
8. International Prognostic Index at low-intermediate, intermediate-high, high risk (2/3/4-5)
9. Adequate haematological counts: ANC > 1.5 x 109/L and platelet count > 75 x 109/L unless due to bone marrow involvement
10. Conjugated bilirubin up to 2 x UNL
11. Alkaline phosphatase and transaminases up to 2 x UNL
12. Creatinine clearance > 50 ml/min
13. HIV negativity
14. HCV negativity
15. HBV negativity or patients with HBVcAb +, HbsAg -, HBs Ab+/- with HBV-DNA negative
16. Cardiac ejection fraction (MUGA scan or echocardiography) > 45%
17. Non peripheral neuropathy or CNS disease. Non testicular Lymphoma
18. Life expectancy > 6 months
19. Performance status < 2 according to ECOG scale
20. Comprehensive geriatric assessment (CGA) as outlined in Appendix 15 showing absence of any impairment in activity of daily living (ADL), of any condition defining a geriatric syndrome, and of any grade 4 comorbidity or of more than three grade 3 comorbidities according to CIRS-G scale
21. Disease free of prior malignancies for ≥ 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
22. Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: for at least 28 days before starting study drug;while participating in the study; for at least 28 days after discontinuation from the study

    * The two methods of reliable contraception must include one highly effective method (i.e., intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e., latex condom, diaphragm, cervical cap)
    * FCBP must be referred to a qualified provider of contraceptive methods if needed

Exclusion Criteria:

1. Lymphoblastic Lymphoma
2. Burkitt Lymphoma
3. Non Hodgkin lymphoma CD 20 negative
4. Mantle Cell Lymphoma
5. Follicular Non Hodgkin Lymphoma grade I-II-IIIa
6. Primitive mediastinal diffuse large B cell lymphoma with only mediastinal involvement
7. International Prognostic Index at low risk (1)
8. Has known or suspected hypersensitivity or intolerance to Rituximab
9. History of evolutive malignancy within the last 3 years other than squamous cell and basal cell carcinoma of the skin or carcinoma in situ of the cervix or breast
10. Extensive radiation therapy, systemic chemotherapy, or other antineoplastic therapy before enrollment within 3 years before the start of treatment
11. Exposure to Rituximab prior to study entry
12. Have received an experimental drug or used an experimental medical device within 4 weeks before the planned start of treatment. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study
13. CNS disease (meningeal and/or brain involvement by lymphoma) or Testicular involvement
14. DVT in the last year
15. History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
16. Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before first dose of study drug
17. Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure (Attachment 5, NYHA Classification of Cardiac Disease), uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
18. Creatinine clearance < 50 ml/min
19. Presence of major neurological disorders
20. HIV positivity
21. HBV positivity with the exception of patients with HBVcAb +, HbsAg -, HBs Ab+/- with HBV-DNA negative
22. HCV positivity
23. Active opportunistic infection
24. Comprehensive geriatric assessment (CGA) as outlined in Appendix 15 showing presence of any impairment in activity of daily living (ADL), of any condition defining a geriatric syndrome, and of any grade 4 comorbidity or of more than three grade 3 comorbidities according to CIRS-G scale
25. Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of adverse events according with Common Terminology Criteria for Adverse events (CTCAE) | 2 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Vitolo, MD, Study Director — Azienda Sanitaria Ospedaliera-Universitaria S. Giovanni Battista - TORINO
Locations (18):
- Italy (18):
  - Divisione di Ematologia Osp. SS. Antonio e Biagio, Alessandria
  - Divisione di Oncologia Medica A Centro di Riferimento Oncologico, Aviano
  - Cattedra di Ematologia Università Policlinico, Bari
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Istituto di Ematologia "Seragnoli" Polic.S.Orsola-Malpighi, Bologna
  - Divisione di Ematologia Spedali Civili, Brescia
  - Divisione di Ematologia Osp. Businco, Cagliari
  - Onco-Ematologia I.R.C.C., Candiolo (TO)
  - Ematologia 1 Ospedale S. Martino, Genova
  - Divisione di Ematologia Ospedale Niguarda, Milan
  - UO Ematologia II Facoltà di Medicina e Chirurgia Università Federico II, Napoli
  - Divisione di Ematologia Università Avogadro, Novara
  - UO Ematologia Università - Policlinico San Matteo, Pavia
  - Dipartimento di biotecnologie cellulari ed ematologia Ospedale Umberto I - La Sapienza, Roma
  - Oncoematologia - Univ. Perugia Sede Terni,, Terni
  - S.C.Ematologia 1 AOU San Giovanni Battista, Torino
  - SC Ematologia 2 ASO San Giovanni Battista, Torino
  - UO Ematologia Osp. Cardinale Panico, Tricase (LE)

REFERENCES:
- [Derived] Vitolo U, Chiappella A, Franceschetti S, Carella AM, Baldi I, Inghirami G, Spina M, Pavone V, Ladetto M, Liberati AM, Molinari AL, Zinzani P, Salvi F, Fattori PP, Zaccaria A, Dreyling M, Botto B, Castellino A, Congiu A, Gaudiano M, Zanni M, Ciccone G, Gaidano G, Rossi G; Fondazione Italiana Linfomi. Lenalidomide plus R-CHOP21 in elderly patients with untreated diffuse large B-cell lymphoma: results of the REAL07 open-label, multicentre, phase 2 trial. Lancet Oncol. 2014 Jun;15(7):730-7. doi: 10.1016/S1470-2045(14)70191-3. Epub 2014 May 13. PMID 24831981
- [Derived] Vose JM, Habermann TM, Czuczman MS, Zinzani PL, Reeder CB, Tuscano JM, Lossos IS, Li J, Pietronigro D, Witzig TE. Single-agent lenalidomide is active in patients with relapsed or refractory aggressive non-Hodgkin lymphoma who received prior stem cell transplantation. Br J Haematol. 2013 Sep;162(5):639-47. doi: 10.1111/bjh.12449. Epub 2013 Jul 9. PMID 23834234
- [Derived] Chiappella A, Tucci A, Castellino A, Pavone V, Baldi I, Carella AM, Orsucci L, Zanni M, Salvi F, Liberati AM, Gaidano G, Bottelli C, Rossini B, Perticone S, De Masi P, Ladetto M, Ciccone G, Palumbo A, Rossi G, Vitolo U; Fondazione Italiana Linfomi. Lenalidomide plus cyclophosphamide, doxorubicin, vincristine, prednisone and rituximab is safe and effective in untreated, elderly patients with diffuse large B-cell lymphoma: a phase I study by the Fondazione Italiana Linfomi. Haematologica. 2013 Nov;98(11):1732-8. doi: 10.3324/haematol.2013.085134. Epub 2013 Jun 28. PMID 23812930